CLINICAL TRIAL: NCT04535544
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-Controlled Study With Deferred Active Treatment to Investigate the Efficacy, Safety, and Pharmacokinetics of JNJ-73763989 + Nucleos(t)Ide Analog in Participants Co-Infected With Hepatitis B and Hepatitis D Virus
Brief Title: A Study of JNJ-73763989 + Nucleos(t)Ide Analog in Participants Co-Infected With Hepatitis B and Hepatitis D Virus
Acronym: REEF-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108868; 2020-001249-37 (EudraCT Number); 73763989HPB2004 (Other: Janssen Research & Development, LLC); 2023-506763-33-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Hepatitis D, Chronic
MeSH Terms: conditions — Hepatitis D, Chronic | interventions — entecavir; Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Immediate Active Treatment arm: JNJ-73763989 + NA (Experimental): Participants will receive JNJ-73763989 subcutaneous (SC) injection every 4 weeks (Q4W) along with NA (entecavir [ETV], tenofovir disoproxil, or tenofovir alafenamide [TAF]) once daily for 144 Weeks in Part 1 and for at least 96 weeks in Part 2.
  Interventions: Drug: JNJ-73763989; Drug: Entecavir (ETV) monohydrate; Drug: Tenofovir disoproxil; Drug: Tenofovir alafenamide (TAF)
- Deferred Active Treatment arm: Placebo+NA+JNJ-73763989+NA (Placebo Comparator): Participants will receive matching placebo to JNJ-73763989 SC injection Q4W along with NA (ETV, tenofovir disoproxil, or TAF) once daily for 52 Weeks followed by JNJ-73763989 SC injection Q4W along with NA once daily for 96 weeks in Part 1 and for at least 48 weeks in Part 2.
  Interventions: Drug: JNJ-73763989; Drug: Placebo; Drug: Entecavir (ETV) monohydrate; Drug: Tenofovir disoproxil; Drug: Tenofovir alafenamide (TAF)

INTERVENTIONS:
Drug: JNJ-73763989 — JNJ-73763989 will be administered as a SC injection.
  Other Names: JNJ-3989
Drug: Placebo — Matching placebo to JNJ-73763989 will be administered as a SC injection.
  Arms: Deferred Active Treatment arm: Placebo+NA+JNJ-73763989+NA
Drug: Entecavir (ETV) monohydrate — ETV monohydrate film coated tablet will be administered orally.
Drug: Tenofovir disoproxil — Tenofovir disoproxil film-coated tablet will be administered orally.
Drug: Tenofovir alafenamide (TAF) — TAF film coated tablet will be administered orally.

SUMMARY:
The purpose of the study is to evaluate on-treatment efficacy against hepatitis D virus (HDV) of JNJ-73763989 + nucleos(t)ide analog (NA) regimen compared to NA alone.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable based on physical examination, medical history, vital signs, electrocardiogram (ECG) at screening
* Chronic hepatitis B virus (HBV) and hepatitis D virus (HDV) co-infection with documentation at least 6 months prior to screening
* For Part 1: hepatitis D RNA (HDV RNA) greater than or equal to (>=) 1000 international units per milliliter (IU/mL) at screening. For Part 2: must have HDV RNA values >= 500 IU/mL, and must have hepatitis B surface antigen (HBsAg) values less than or equal to (<=) 10000 IU/mL at screening or HDV RNA values at screening are <= 100000 IU/mL
* Alanine aminotransferase (ALT) greater than upper limit normal (ULN) but less than 10 times (ULN)
* Body mass index (BMI) between 18.0 and 35.0 kilogram per meter square (kg/m^2), extremes included
* Highly effective contraceptive measures in place for female participants of childbearing potential or male participants with female partners of childbearing potential
* Non-cirrhotic participants and participants with compensated cirrhosis (Child Pugh class A) at screening (Part 1) and participants must have absence of cirrhosis and platelet count of >= 140000 per deciliter (dL) for enrollment into Part-2

Exclusion Criteria:

* Evidence of infection with hepatitis A, C, or E virus infection or evidence of human immunodeficiency, virus type 1 (HIV-1) or HIV-2 infection at screening
* History or evidence of clinical signs/symptoms of hepatic decompensation including but not limited to: portal hypertension, ascites, hepatic encephalopathy, esophageal varices or any laboratory abnormalities indicating a reduced liver function as defined in the protocol
* Evidence of liver disease of non-HBV/HDV etiology
* Signs of hepatocellular carcinoma (HCC)
* Significant laboratory abnormalities as defined in the protocol at screening
* Participants with a history of malignancy within 5 years before screening
* Abnormal sinus rhythm or ECG parameters at screening as defined in the protocol
* History of or current cardiac arrhythmia or history or clinical evidence of significant or unstable cardiac disease
* Participants with any current or previous illness for which, in the opinion of the investigator and/or sponsor, participation would not be in the best interest of the participant
* History of or current clinically significant skin disease or drug rash
* Participants with known allergies, hypersensitivity, or intolerance to JNJ-3989 or its excipients or excipients of the placebo content
* Contraindications to the use of entecavir (ETV), tenofovir disoproxil, or tenofovir alafenamide (TAF) per local prescribing information
* Participants who have taken any therapies disallowed per protocol
* Female participants who are pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 90 days after the last dose of study intervention
* Male participants who plan to father a child while enrolled
* Participants who had or planned major surgery, (example, requiring general anesthesia) or who have received an organ transplant
* Vulnerable participants (example, incarcerated individuals, individuals under a legal protection measure)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2025-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (61):
- United States (2):
  - Stanford University School of Medicine, Redwood City, California
  - Harvard Medical School Massachusetts General Hospital, Boston, Massachusetts
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown
  - Western Health, Footscray
  - Westmead Hospital, Westmead
- Brazil (3):
  - Centro Oncológico De Roraima, Boa Vista
  - Fundacao De Medicina Tropical Doutor Heitor Vieira Dourado, Manaus
  - Cepem - Centro de Pesquisa Em Medicina Tropical, Porto Velho
- China (9):
  - Beijing Ditan Hospital Capical Medical University, Beijing
  - Peking University People s Hospital, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - West China Hospital Sichuan University, Chengdu
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Guangzhou Eighth People's Hospital, Guangzhou Medical University, Guangzhou
  - Nanfang Hospital, Guangzhou
  - The First Affiliated Hospital Zhejiang University College of Medicine, Hangzhou
  - Huashan Hospital Fudan University, Shanghai
- France (5):
  - Hopital Beaujon, Clichy
  - Hopital de La Croix Rousse, Lyon
  - CHU de Nantes hotel Dieu, Nantes
  - CHU Hopital Saint Antoine, Paris
  - Chu Rennes Hopital Pontchaillou, Rennes
- Germany (3):
  - Universitatsklinikum Essen, Essen
  - Universitätsklinikum Johann Wolfgang Goethe- Universität Frankfurt Medizinische Klinik 1, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
- Italy (4):
  - Irccs Ospedale Maggiore Di Milano, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Universita degli Studi di Roma 'La Sapienza' - Umberto I Policlinico di Roma, Rome
  - Ospedale Molinette, AO Città della Salute e della Scienza di, Torino
- Japan (13):
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - National Hospital Organization Shikoku Cancer Center, Iizuka-shi
  - Ikeda City Hospital, Ikeda
  - Kumamoto University Hospital, Kumamoto
  - Kumamoto Shinto General Hospital, Kumamoto
  - Nagasaki University Hospital, Nagasaki
  - National Hospital Organization Nagasaki Medical Center, Nagasaki
  - University of the Ryukyus Hospital, Nakagami Gun
  - Nakagami Hospital, Okinawa
  - Suita Municipal Hospital, Suita
  - Osaka University Hospital, Suita-shi
  - Tokyo Metropolitan Bokutoh Hospital, Sumida Ku
- New Zealand Clinical Research, Auckland, New Zealand
- Russia (3):
  - Krasnoyarsk Regional Center For AIDS And Infectious Diseases Treatment And Prophylaxis, Krasnoyarsk
  - St. Petersburg City Center for AIDS and Infectious Diseases Treatment and Prophylaxis, Saint Petersburg
  - Medical Company Hepatolog Ltd, Samara
- Spain (4):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. Marques de Valdecilla, Santander
- Sweden (3):
  - Danderyds Sjukhus, Danderyd
  - Skanes universitetssjukhus, Malmo
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
- Taiwan (3):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - China Medical University Hospital, Tiachung
- Turkey (Türkiye) (4):
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Ege University Medical of Faculty, Department of Gastroenterology, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Karadeniz Teknik University Medical Faculty, Trabzon
- Kings College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants co-infected with hepatitis B virus (HBV) and hepatitis D virus (HDV) were considered eligible for participation. Participants with compensated cirrhosis were allowed to be enrolled in Part 1 but excluded from Part 2 of the study.
Pre-assignment Details: The study consisted of 2 parts: 1 and 2. Part 2 was initiated when the protocol specified antiviral activity criteria was met in Part 1 and when all participants of Part 1 had completed at least Week 16 or discontinued earlier. Unique participants were randomized (4:1) to JNJ-73763989 + NA and Placebo + NA in Part 1 and 2. Two ongoing participants in double-blind phase Part 2 completed Week 48 visit. Hence, included in the primary analysis at Week 48.
Groups:
- Part 1: JNJ-73763989 + Nucleos(t)Ide Analog (NA): In the double-blind phase, participants received JNJ-73763989 100 milligrams (mg) subcutaneous (SC) injection every 4 weeks (Q4W) along with NA (entecavir [ETV] monohydrate 0.5 mg, tenofovir disoproxil 245 mg, or tenofovir alafenamide [TAF] 25 mg) tablet orally once daily for 52 weeks. After completion of double-blind phase, participants entered open-label phase and continued to receive JNJ-73763989 100 mg SC injection Q4W along with NA (ETV 0.5 mg, tenofovir disoproxil 245 mg, or TAF 25 mg) tablet orally once daily for 92 weeks (up to Week 144). After completion of open-label phase, participants entered 48-week follow-up phase during which JNJ-73633989 treatment was stopped and NA treatment alone was continued.
- Part 1: Placebo + NA: In the double-blind phase, participants received placebo matching to JNJ-73763989 SC injection Q4W along with NA (ETV 0.5 mg, tenofovir disoproxil 245 mg, or TAF 25 mg) tablet orally once daily for 52 weeks. After completion of double-blind phase, participants entered open-label phase and received JNJ-73763989 100 mg SC injection Q4W along with NA (ETV 0.5 mg, tenofovir disoproxil 245 mg, or TAF 25 mg) tablet orally once daily for 96 weeks (up to Week 148). After completion of open-label phase, participants entered 48-week follow-up phase during which JNJ-73633989 treatment was stopped and NA treatment alone was continued.
- Part 2: JNJ-73763989 + NA: In the double-blind phase, participants received JNJ-73763989 100 mg SC injection Q4W along with NA (ETV 0.5 mg, tenofovir disoproxil 245 mg, or TAF 25 mg) tablet orally once daily for 52 weeks. After completion of double-blind phase, participants entered open-label phase and continued to receive JNJ-73763989 100 mg SC injection Q4W along with NA (ETV 0.5 mg, tenofovir disoproxil 245 mg, or TAF 25 mg) tablet orally once daily for 92 weeks (up to Week 144). After completion of open-label phase, participants entered 48-week follow-up phase and stopped JNJ-73633989 treatment and continued NA treatment alone.
- Part 2: Placebo + NA: In the double-blind phase, participants received placebo matching to JNJ-73763989 SC injection Q4W along with NA (ETV 0.5 mg, tenofovir disoproxil 245 mg, or TAF 25 mg) tablet orally once daily for 52 weeks. After completion of double-blind phase, participants entered open-label phase and received JNJ-73763989 100 mg SC injection Q4W along with NA (ETV 0.5 mg, tenofovir disoproxil 245 mg, or TAF 25 mg) tablet orally once daily for 96 weeks (up to Week 148). After completion of open-label phase, participants entered 48-week follow-up phase and stopped JNJ-73633989 treatment and continued NA treatment alone.
Period: Double-blind (Day 1 up to Week 52)
Arm/Group | Part 1: JNJ-73763989 + Nucleos(t)Ide Analog (NA) | Part 1: Placebo + NA | Part 2: JNJ-73763989 + NA | Part 2: Placebo + NA
Started | 17 | 5 | 24 | 6
Completed | 16 | 5 | 20 | 5
Not Completed | 1 | 0 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 0
Not completed — Ongoing after Week 48 | 0 | 0 | 1 | 1
Period: Open-label (Week 52 up to Week 148)
Arm/Group | Part 1: JNJ-73763989 + Nucleos(t)Ide Analog (NA) | Part 1: Placebo + NA | Part 2: JNJ-73763989 + NA | Part 2: Placebo + NA
Started | 5 (11 participants who discontinued treatment with JNJ-73763989 during the double-blind phase, completed the end of treatment visit and moved directly to follow-up without entering the open label phase.) | 4 (1 participant who discontinued treatment with JNJ-73763989 during the double-blind phase, completed the end of treatment visit and moved directly to follow-up without entering the open label phase.) | 14 (6 participants who discontinued treatment with JNJ-73763989 during the double-blind phase, completed the end of treatment visit and moved directly to follow-up without entering the open label phase.) | 5
Completed | 5 | 2 | 0 | 0
Not Completed | 0 | 2 | 14 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Ongoing | 0 | 1 | 14 | 4
Period: Follow-up (Week 148 up to Week 161)
Arm/Group | Part 1: JNJ-73763989 + Nucleos(t)Ide Analog (NA) | Part 1: Placebo + NA | Part 2: JNJ-73763989 + NA | Part 2: Placebo + NA
Started | 16 (5 participants who completed open-label phase + 11 participants who discontinued treatment with JNJ-73763989 during the double-blind phase, completed the end of treatment visit and moved directly to follow-up without entering the open label phase.) | 3 (2 participants who completed open-label phase + 1 participant who discontinued treatment with JNJ-73763989 during the double-blind phase, completed the end of treatment visit and moved directly to follow-up without entering the open label phase.) | 6 (6 participants who discontinued treatment with JNJ-73763989 during the double-blind phase, completed the end of treatment visit and moved directly to follow-up without entering the open label phase.) | 0
Completed | 7 | 3 | 1 | 0
Not Completed | 9 | 0 | 5 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 4 | 0
Not completed — Ongoing | 4 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: JNJ-73763989 + Nucleos(t)Ide Analog (NA) | Part 1: Placebo + NA | Part 2: JNJ-73763989 + NA | Part 2: Placebo + NA | Total
Number analyzed (Participants) | 17 | 5 | 24 | 6 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 5 | 24 | 6 | 52
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (10.44) | 44.2 (11.88) | 43.8 (9.49) | 44.8 (11.96) | 43 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 9 | 3 | 23
  Male | 9 | 2 | 15 | 3 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 15 | 5 | 24 | 6 | 50
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 0 | 4
  Black or African American | 1 | 0 | 2 | 1 | 4
  White | 13 | 4 | 20 | 4 | 41
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  FRANCE | 0 | 0 | 2 | 0 | 2
  GERMANY | 0 | 0 | 1 | 1 | 2
  ITALY | 0 | 0 | 8 | 2 | 10
  NEW ZEALAND | 4 | 1 | 1 | 0 | 6
  RUSSIAN FEDERATION | 3 | 0 | 0 | 0 | 3
  SPAIN | 3 | 0 | 1 | 0 | 4
  SWEDEN | 1 | 0 | 1 | 0 | 2
  TAIWAN | 0 | 0 | 0 | 1 | 1
  TURKEY | 2 | 4 | 8 | 1 | 15
  UNITED KINGDOM | 3 | 0 | 1 | 1 | 5
  UNITED STATES | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Double-blind: Part 1: Percentage of Participants With HDV Ribonucleic Acid (RNA) >=2 log10 IU/mL Decline From Baseline or HDV RNA Target Not Detected (TND) in Combination With Normal Alanine Aminotransferase (ALT) at Week 48 (Multiple Imputation Approach)
Description: Percentage of participants with HDV RNA greater than or equal to (>=) 2 log10 International Units Per Milliliter (IU/mL) decline from baseline or HDV RNA TND in combination with normal ALT at Week 48 using multiple imputation approach was reported. Target not detected (TND) was defined as no traces of HBV RNA were detected/found. Normal ALT was defined as ALT less than (<) upper limit of normal (ULN) with ULN = 34 units per liter (U/L) for female and 43 U/L for male. The baseline assessment was defined as the last observed non-missing measurement before the date and time of the first administration of any of study intervention on Day 1. The multiple imputation approach was derived using a longitudinal multiple regression model to impute missing data.
Time Frame: At Week 48
Population: Intent-to-Treat analysis set (ITT) included all participants who were randomly assigned to an intervention arm and who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they were randomly assigned to.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: JNJ-73763989 + Nucleos(t)Ide Analog (NA) | Part 1: Placebo + NA
Number analyzed (Participants) | 17 | 5
Percentage of Participants | 23.5 | 0.0
Statistical Analysis 1: Comparison: Part 1: JNJ-73763989 + Nucleos(t)Ide Analog (NA) vs Part 1: Placebo + NA; Stratum-adjusted Mantel-Haenszel (MH) test was used to assess the difference of percentage based on stratification factor: HBeAg status at screening (positive vs negative); Test type: Superiority; p = 0.011, Mantel-Haenszel; Difference of percentage = 23.7, 95% CI 2-sided [3.52 to 43.96]

2. Primary Outcome: Double-blind: Part 2: Percentage of Participants With HDV RNA >=2 log10 IU/mL Decline From Baseline or HDV RNA TND in Combination With ALT at Week 48 (Multiple Imputation Approach)
Description: Percentage of participants with HDV RNA >=2 log10 IU/mL decline from baseline or HDV RNA TND in combination with normal ALT at Week 48 using multiple imputation approach was reported. TND was defined as no traces of HBV RNA were detected/found. Normal ALT was defined as ALT <ULN with ULN = 34 U/L for female and 43 U/L for male. The baseline assessment was defined as the last observed non-missing measurement before the date and time of the first administration of any of study intervention on Day 1. The multiple imputation approach was derived using a longitudinal multiple regression model to impute missing data.
Time Frame: At Week 48
Population: ITT analysis set included all participants who were randomly assigned to an intervention arm and who received at least 1 dose of study intervention. Participants were analyzed according to the study intervention they were randomly assigned to.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2: JNJ-73763989 + NA | Part 2: Placebo + NA
Number analyzed (Participants) | 24 | 6
Percentage of Participants | 27.1 | 0.0
Statistical Analysis 1: Comparison: Part 2: JNJ-73763989 + NA vs Part 2: Placebo + NA; Stratum-adjusted MH test was used to assess the difference of percentage based on stratification factor: HBeAg status at screening (positive vs negative); Test type: Superiority; p = 0.003, Mantel-Haenszel; Difference of percentage = 26.8, 95% CI 2-sided [7.38 to 46.21]

ADVERSE EVENTS:
Time Frame: From Day 1 to Week 52 in double-blind (DB) phase, from Week 52 to Week 148 in open-label (OL) phase and from Week 148 to Week 161 in follow-up (FU) phase
Description: Safety analysis set included all participants who took at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received. Adverse event data collection is still ongoing and will be updated upon study completion. As none of the participants entered the follow-up phase from open-label phase 'Part 2: Placebo + NA' arm, hence, no data was collected and this arm is not reported in adverse event section.
Groups:
- DB: Part 1: JNJ-73763989 + NA; DB: Part 2: JNJ-73763989 + NA: In the double-blind phase, participants received JNJ-73763989 100 mg SC injection Q4W along with NA (ETV 0.5 mg, tenofovir disoproxil 245 mg, or TAF 25 mg) tablet orally once daily for 52 weeks.
- DB: Part 1: Placebo + NA; DB: Part 2: Placebo + NA: In the double-blind phase, participants received placebo matching to JNJ-73763989 SC injection Q4W along with NA (ETV 0.5 mg, tenofovir disoproxil 245 mg, or TAF 25 mg) tablet orally once daily for 52 weeks.
- OL: Part 1: JNJ-73763989 + NA; OL: Part 2: JNJ-73763989 + NA: After completion of double-blind phase, participants entered open-label phase and continued to receive JNJ-73763989 100 mg SC injection Q4W along with NA (ETV 0.5 mg, tenofovir disoproxil 245 mg, or TAF 25 mg) tablet orally once daily for 92 weeks (up to study Week 144).
- OL: Part 1: Placebo + NA; OL: Part 2: Placebo + NA: After completion of double-blind phase, participants entered open-label phase and received JNJ-73763989 100 mg SC injection Q4W along with NA (ETV 0.5 mg, tenofovir disoproxil 245 mg, or TAF 25 mg) tablet orally once daily for 96 weeks (up to study Week 148).
- FU: Part 1: JNJ-73763989 + NA; FU: Part 1: Placebo + NA: After completion of open-label phase, participants entered 48-week follow-up phase during which JNJ-73633989 treatment was stopped and NA treatment alone was continued.
- FU: Part 2: JNJ-73763989 + NA: After completion of open-label phase, participants entered 48-week follow-up phase and stopped JNJ-73633989 treatment and continued NA treatment alone.
Arm/Group | DB: Part 1: JNJ-73763989 + NA | DB: Part 1: Placebo + NA | DB: Part 2: JNJ-73763989 + NA | DB: Part 2: Placebo + NA | OL: Part 1: JNJ-73763989 + NA | OL: Part 1: Placebo + NA | OL: Part 2: JNJ-73763989 + NA | OL: Part 2: Placebo + NA | FU: Part 1: JNJ-73763989 + NA | FU: Part 1: Placebo + NA | FU: Part 2: JNJ-73763989 + NA
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/5 | 0/24 | 0/6 | 0/5 | 0/4 | 0/14 | 0/5 | 0/16 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/17 | 0/5 | 3/24 | 0/6 | 0/5 | 1/4 | 0/14 | 0/5 | 1/16 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 17/17 | 3/5 | 20/24 | 5/6 | 4/5 | 4/4 | 2/14 | 2/5 | 11/16 | 3/3 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Part 1: JNJ-73763989 + NA (N=17) | DB: Part 1: Placebo + NA (N=5) | DB: Part 2: JNJ-73763989 + NA (N=24) | DB: Part 2: Placebo + NA (N=6) | OL: Part 1: JNJ-73763989 + NA (N=5) | OL: Part 1: Placebo + NA (N=4) | OL: Part 2: JNJ-73763989 + NA (N=14) | OL: Part 2: Placebo + NA (N=5) | FU: Part 1: JNJ-73763989 + NA (N=16) | FU: Part 1: Placebo + NA (N=3) | FU: Part 2: JNJ-73763989 + NA (N=6)
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intermenstrual Bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Part 1: JNJ-73763989 + NA (N=17) | DB: Part 1: Placebo + NA (N=5) | DB: Part 2: JNJ-73763989 + NA (N=24) | DB: Part 2: Placebo + NA (N=6) | OL: Part 1: JNJ-73763989 + NA (N=5) | OL: Part 1: Placebo + NA (N=4) | OL: Part 2: JNJ-73763989 + NA (N=14) | OL: Part 2: Placebo + NA (N=5) | FU: Part 1: JNJ-73763989 + NA (N=16) | FU: Part 1: Placebo + NA (N=3) | FU: Part 2: JNJ-73763989 + NA (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Motion Sickness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis Allergic (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Varices Oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling Hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Discolouration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel Puncture Site Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Autoimmune Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gallbladder Polyp (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic Fibrosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteriuria (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth Abscess (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb Crushing Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Nausea (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 9 | 0 | 7 | 1 | 1 | 2 | 0 | 0 | 3 | 1 | 4
Amylase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 7 | 0 | 4 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 2
Beta 2 Microglobulin Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bilirubin Conjugated Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Bilirubin Increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Human Chorionic Gonadotropin Positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver Function Test Abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases Increased (Investigations) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma of Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Burning Sensation (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intercostal Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Trigeminal Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depressed Mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia Areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulite (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT04535544/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT04535544/SAP_001.pdf